CLINICAL TRIAL: NCT00500864
Title: Effects of Acute Intravenous Magnesium Loading on Pulmonary Function Parameters and Maximal Exercise Capacity of Patients With Chronic Obstructive Pulmonary Disease in Stable Clinical Conditions.
Brief Title: Magnesium Loading in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HCFMRP8518/2003
Record Dates: First submitted 2007-07-12; First posted 2007-07-13 (Estimated); Last update posted 2008-07-02 (Estimated); Status verified 2008-06

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Magnesium; Pulmonary function; Exercise Physiology
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Magnesium Sulfate 2 grams

SUMMARY:
Dietary magnesium (Mg) intake has been shown to be independently related to lung function, airway reactivity, and respiratory symptoms in the general population. Inhaled Mg and IV Mg administration have been shown to promote bronchodilation and to improve lung function in asthmatic patients. Some studies have suggested that COPD patients exhibit decreased body levels of Mg. The purpose of the present study was to investigate the effects of acute IV Mg loading on parameters of respiratory function and maximal exercise capacity of stable COPD patients.The study hypothesis is that Mg administration will be associated to improvements on airflow and vasodilation leading to improvements of pulmonary function and exercise performance.

DETAILED DESCRIPTION:
Patients are required to have a diagnosis of COPD according to the Global Initiative for Chronic Obstructive Lung Disease criteria.

This is a randomized, double-blind, placebo-controlled, cross-over study. Twenty five patients are going to be included. They are going to come to the laboratory to receive IV placebo or IV Mg sulfate at two distinct occasions about 48 hours apart. Half of the patients are going to receive Mg first and Placebo at the second day, while the other half are going to receive the treatments in an inverse order. Tests are going to be performed before and about 40 minutes after the IV infusions. Tests to be performed are: spirometry, arterial blood gases, Mg plasma level measurements, and a maximal exercise test protocol in cycloergometer.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis according GOLD criteria
* Men between 45 and 80 years old

Exclusion Criteria:

* History of asthma or atopy, renal failure, heart failure, arrhythmias or cardiac electrical disturbances, and other significant disease other than COPD.
* Individuals on chronic oral steroids, diuretics, or use of mineral supplementation.
* Locomotor impairment.

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-08; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Measurements of forced vital capacity (FVC), forced expiratory volume (FEV1), functional residual capacity (FRC),maximal respiratory pressures,maximal oxygen consumption and maximal work load. | Immediatly after the end of IV infusion

SECONDARY OUTCOMES:
Arterial blood gases at rest, heart rate and mean arterial blood pressure. Degree of desaturation during maximal exercise. | Immediatly after the end of IV infusion

CONTACTS AND LOCATIONS:
Overall Officials: José B Martinez, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clínicas de Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Derived] Amaral AF, Gallo L Jr, Vannucchi H, Crescencio JC, Vianna EO, Martinez JA. The effect of acute magnesium loading on the maximal exercise performance of stable chronic obstructive pulmonary disease patients. Clinics (Sao Paulo). 2012;67(6):615-22. doi: 10.6061/clinics/2012(06)12. PMID 22760901